CLINICAL TRIAL: NCT02293707
Title: A Randomised, Parallel-group, Open-label Phase II Trial of the Immunological Effects of Three Regimens of GX301 Vaccination in Castration-resistant Prostate Cancer Patients Who Have Achieved Response or Disease Stability With First-line Chemotherapy
Brief Title: A Phase II Randomised Trial of Three Regimens of GX301 Vaccination in Castration-resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratoires Leurquin Mediolanum (Industry)
Collaborators: Universita degli Studi di Genova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MED-GX301-02; 2014-000095-26 (EudraCT Number)
Record Dates: First submitted 2014-11-14; First posted 2014-11-18 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer
Keywords: Castration-resistant prostate cancer; Therapeutic vaccine; Telomerase vaccine
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GX301 Regimen A (8 administrations) (Experimental): Administration time frame: Day 1 to Day 63.
  Interventions: Biological: GX301
- GX301 Regimen B (4 administrations) (Experimental): Administration time frame: Day 1 to Day 63.
  Interventions: Biological: GX301
- GX301 Regimen C (2 administrations) (Experimental): Administration time frame: Day 1 to Day 63.
  Interventions: Biological: GX301

INTERVENTIONS:
Biological: GX301 — GX301 therapy consists of four human telomerase reverse transcriptase (hTERT) peptides and two adjuvants.
  Peptides are hTERT (540-548) Acetate, hTERT (611-626) Acetate, hTERT (672-686) Acetate and hTERT (766-780) Acetate. Adjuvants are Montanide ISA 51 VG and imiquimod 5% cream (Aldara).
  Each GX301 administration will consist of four intradermal injections - one injection for each hTERT peptide - given at the same time and followed by topical application of imiquimod. Each intradermal injection will consist of a fixed hTERT peptide dose, 500 µg, reconstituted as a solution and mixed with Montanide ISA 51 VG.

SUMMARY:
GX301 is an experimental therapeutic vaccine directed against human telomerase, an enzyme playing an essential role in cancer cell proliferation.

This clinical trial will test three different GX301 administration regimens in castration-resistant prostate cancer patients who have achieved response or disease stability with first-line docetaxel treatment. This is aimed at identifying an optimal vaccination regimen.

The three regimens will primarily be compared for their efficacy and safety in inducing vaccine-specific immunological responses over a period of 6 months following treatment initiation. In addition, patients will be observed for the occurrence of disease progression and for their vital status up to 24 months.

DETAILED DESCRIPTION:
GX301, an experimental therapeutic (anti-cancer) vaccine, is composed of four immunogenic peptides from human telomerase and two complementary adjuvants, Montanide ISA-51 VG and imiquimod.

An earlier Phase 1 study of GX301 has provided evidence of vaccine-specific immune response in a small sample of stage 4 prostate cancer patients given eight GX301 administrations over 9 weeks.

The present Phase 2, randomised, parallel-group, multicentre trial is aimed at comparing three different GX301 administration regimens in patients with progressive, castration-resistant prostate cancer who have completed a first-line docetaxel treatment and have achieved response to chemotherapy or disease stability. Primary comparisons will include regimen efficacy in inducing vaccine-specific immunological responses over a period of 6 months following randomisation; and treatment safety and tolerability over the same period.

A further study aim is to investigate whether achievement of immunological response, irrespective of the assigned GX301 regimen, is related to progression-free and/or overall survival.

Eligible patients will be randomly assigned to receive one of three GX301 vaccination regimens consisting of two, four or eight administrations, respectively, each regimen being given over a fixed 9-week period. Randomisation ratio will be 1:1:1. Randomisation will be stratified by previous cumulative exposure to docetaxel.

Following randomisation, immunological responses to GX301 will be determined over a 6-month period. However, on-study patient observation will be continued until the occurrence of one of the following end-points, whichever the earliest: (a) disease progression; (b) death; (c) completion of an 18-month observation period; or (d) patient's decision to terminate his participation in the study.

All patients discharged from the trial for reasons (a) or (c) will undergo a follow-up to ascertain survival until 24 months from randomisation.

Data analysis will be carried out in two sequential steps. The first step will focus on co-primary outcomes and will therefore take place upon completion of the study dataset up to the 6-month time-point. The second step will incorporate secondary outcomes and will therefore be conducted upon completion of the full study dataset.

ELIGIBILITY:
Inclusion Criteria:

Documented patient history

* Histologically confirmed diagnosis of prostate cancer, with an available Gleason score.
* Diagnosis of progressive, castration-resistant prostate cancer (CRPC), leading to inception of first-line chemotherapy with a docetaxel-based regimen.
* Completion of chemotherapy with a cumulative delivered dose of 300 to 825 mg/m2 docetaxel.

Note: Pre-chemotherapy exposure to abiraterone and prednisone does not preclude eligibility, provided that both agents have been discontinued prior to initiation of docetaxel.

Current patient status

* Ability to understand study-related patient information and provision of written informed consent for participation in the study.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of at least 6 months.
* An interval ≥4 weeks elapsed from the last docetaxel administration.
* Documented achievement of response or disease stability with docetaxel chemotherapy.
* Absence of cancer-related symptoms suggesting clinical disease progression.
* Current castrate testosterone level (≤50 ng/dL) due to current gonadotropin-releasing hormone (GnRH) agonist or antagonist therapy or past orchiectomy.
* Haematology and blood chemistry tests within specified limits.
* Successful recovery from acute toxicities from prior chemotherapy.
* Confirmation from the immunology laboratory that the blood sample provided for baseline immunological tests is technically adequate.

Exclusion Criteria:

* Known intolerance to Montanide or imiquimod.
* Known presence of brain metastatic disease or spinal cord compression.
* Radiotherapy within the past 4 weeks.
* Concomitant presence of other primary malignancy
* Major surgery within 4 weeks prior to randomisation.
* Cardiovascular illness or complication which, in Investigator's judgment, compromises prognosis at 6 months or prevents the patient from following study procedures.
* Serious uncontrolled infection.
* Known presence of active autoimmune disease.
* Known presence of acquired, hereditary, or congenital immunodeficiency.
* HIV infection.
* Current need for immunosuppressive drug therapy, including systemic corticosteroids.
* Current need for denosumab therapy. (Patients under bisphosphonate treatment are eligible).
* Skin disease interfering with evaluation of local tolerance of GX301 injections.
* Participation in any interventional drug or medical device study within 30 days prior to treatment start.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2014-11; Primary Completion 2018-08 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Achievement of immunological response | Days 90 and 180 following randomisation
Incidence of adverse events | Up to Day 180
Changes from baseline in laboratory tests for immunological safety | Days 63, 90 and 180

SECONDARY OUTCOMES:
Changes from baseline in serum prostate-specific antigen (PSA) | Up to Day 540 or end of observation (if earlier)
Progression-free survival | Up to Day 540 or end of observation (if earlier)
Overall survival | Up to Day 720
Incidence of adverse events | Up to Day 540 or end of observation (if earlier)
Changes from baseline in laboratory tests for immunological safety | Up to Day 540 or end of observation (if earlier)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Boccardo, MD, Principal Investigator — DIMI, Università di Genova - Clinica di Oncologia Medica, IRCCS San Martino-IST
Locations (24):
- Italy (17):
  - S.C. di Oncologia, A.S.O. "Santi Antonio e Biagio e Cesare Arrigo", Alessandria
  - Oncologia Medica A, Centro di Riferimento Oncologico (CRO), Aviano
  - Oncologia Medica, Azienda Ospedaliero Universitaria - Policlinico Consorziale, Bari
  - U.O.C. Urologia 1, A.O.U. Consorziale Policlinico di Bari, Bari
  - Oncologia Medica, A.O. Spedali Civili, Brescia
  - S.C. Oncologia Medica, Presidio Ospedaliero Busto Arsizio, Busto Arsizio
  - IRCCS Fondazione del Piemonte per l'Oncologia (FPO), Candiolo
  - Clinica di Oncologia Medica, IRCCS San Martino-IST, Genova
  - U.O. Medicina Oncologica - Ospedale San Raffaele IRCCS, Milan
  - Unità Oncologica Medica Urogenitale, Istituto Europeo di Oncologia, Milan
  - Dipartimento Uro-Ginecologico, IRCCS Istituto Nazionale Tumori - Fondazione Pascale, Napoli
  - U.O.C. di Oncologia Medica, A.O.R.N. "Antonio Cardarelli", Napoli
  - Oncologia Medica, A.O. Universitaria San Luigi Gonzaga, Orbassano
  - U.O. di Oncologia, AUSL di Piacenza, Piacenza
  - Unita Oncologica, Azienda Ospedaliera S. Maria degli Angeli, Pordenone
  - U.O.C. di Oncologia Medica, Policlinico "Le Scotte", Siena
  - Oncologia Medica d.U., Policlinico G.B. Rossi, A.O.U.I. Verona, Verona
- Spain (7):
  - Medical Oncology, Hospital Vall d'Hebron, Barcelona
  - Hospital Clìnic i Provincial de Barcelona, Barcelona
  - Medical Oncology, Institut Català d'Oncologìa, L'Hospitalet de Llobregat, Barcelona
  - Oncología, Hospital Universitario Gregorio Marañón, Madrid
  - Servicio de Oncologìa Médica, Hospital Universitario Ramòn y Cajal, Madrid
  - Oncología Médica, Hospital Clínico San Carlos, Madrid
  - Oncology, Corporaciò Sanitària Parc Taulì, Sabadell, Barcelona

REFERENCES:
- [Background] Fenoglio D, Traverso P, Parodi A, Tomasello L, Negrini S, Kalli F, Battaglia F, Ferrera F, Sciallero S, Murdaca G, Setti M, Sobrero A, Boccardo F, Cittadini G, Puppo F, Criscuolo D, Carmignani G, Indiveri F, Filaci G. A multi-peptide, dual-adjuvant telomerase vaccine (GX301) is highly immunogenic in patients with prostate and renal cancer. Cancer Immunol Immunother. 2013 Jun;62(6):1041-52. doi: 10.1007/s00262-013-1415-9. Epub 2013 Apr 17. PMID 23591981
- [Background] Fenoglio D, Parodi A, Lavieri R, Kalli F, Ferrera F, Tagliamacco A, Guastalla A, Lamperti MG, Giacomini M, Filaci G. Immunogenicity of GX301 cancer vaccine: Four (telomerase peptides) are better than one. Hum Vaccin Immunother. 2015;11(4):838-50. doi: 10.1080/21645515.2015.1012032. PMID 25714118
- [Derived] Filaci G, Fenoglio D, Nole F, Zanardi E, Tomasello L, Aglietta M, Del Conte G, Carles J, Morales-Barrera R, Guglielmini P, Scagliotti G, Signori A, Parodi A, Kalli F, Astone G, Ferrera F, Altosole T, Lamperti G, Criscuolo D, Gianese F, Boccardo F. Telomerase-based GX301 cancer vaccine in patients with metastatic castration-resistant prostate cancer: a randomized phase II trial. Cancer Immunol Immunother. 2021 Dec;70(12):3679-3692. doi: 10.1007/s00262-021-03024-0. Epub 2021 Aug 5. PMID 34351436